CLINICAL TRIAL: NCT04995796
Title: Testing the Decision Aid: Supporting Patient Decisions About Upper Extremity Surgery in Cervical Spinal Cord Injury (AIM 3)
Brief Title: Testing the Decision Aid: Supporting Patient Decisions About Upper Extremity Surgery in Cervical SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ida Fox, Associate Professor of Surgery, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202106018
Record Dates: First submitted 2021-07-07; First posted 2021-08-09 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Cervical Spinal Cord Injury; Tetraplegia
Keywords: Nerve Transfer Surgery; Tendon Transfer Surgery; Decision Support Intervention
MeSH Terms: conditions — Quadriplegia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Prospective, single arm pre/post pilot study. This non-therapeutic study will provide no direct medical benefit to the research participants but will help the researchers learn more so that future generations may benefit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled Participants (Experimental): Study participation will involve 2 visits. The first visit will take approximately 90 minutes, but may be longer if participant desires longer interaction with the DSI/DA. The second visit will take approximately 5 minutes.
  Interventions: Other: Surveys for Research Purposes

INTERVENTIONS:
Other: Surveys for Research Purposes — VISIT #1:
  1. Pre-Testing:
     * Pre Knowledge Test
     * Pre SURE (decisional conflict) test
  2. Independent DSI/DA Interaction
  3. Post-Testing:
     * Post Knowledge Test
     * Post SURE (decisional conflict) Test
     * Acceptability Index
     * Modified Single Item Literacy Screen
     * Additional Demographics
  VISIT #2: Check-In Call 1 week later:
  After viewing the DSI/DA and completing the post-test components above, the subjects will also complete a 5 minute debrief interview about 1 week later via phone or video conference with a team member to give feedback on their experience using the DSI/DA, including its strengths and weaknesses. This will allow for further improvement and refinement of the DSI.

SUMMARY:
Purpose: The objective of this study is to assess a newly created decision support intervention (DSI) or decision aid (DA) for people with spinal cord injury (SCI) to learn about and consider upper extremity reconstructive surgery to help them choose a course of treatment that most aligns with their values.

DETAILED DESCRIPTION:
The overarching aim of this project is to define key information about improvement of upper extremity function after SCI (time and extent of recovery, outcome of surgical and non-surgical interventions and the experience thereof) and communicate this information to patients and clinicians to support their treatment decisions.

This particular Aim 3 of the overall project will assess a newly developed DSI/DA tool in a pre-/post- pilot study of people with SCI hoping to restore upper extremity function in cervical SCI. Using information from prior aims of this project, a de novo tool has been created and will be tested. This study will measure participant knowledge of their condition and treatment options, and decisional conflict. Participant feedback, demographics, and health-literacy information will be collected to help improve and refine the DA before it is made widely available to the public.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (≥18 years to ≤80 years) with mid-cervical level SCI (minimum 6 months and maximum 20 years post-injury).
2. Must have limited use of their hands.
3. Wheelchair dependent for mobility.
4. Ability to read, speak and understand English.

Exclusion Criteria:

1) Previous treatment with nerve or tendon transfer surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Knowledge Questionnaire | At baseline and then immediately after reviewing the Decision Aid (estimated to be around 60-90 minutes later).
  An online, novel, 10-question knowledge survey will provide information about the Decision Aid's effect on patient understanding of their condition, treatment options, and probability of recovery. This questionnaire will be administered as a "Pre-Test" before participants view the Decision Aid, and then later as a "Post-Test" after participants view the Decision Aid.
  Hypothesis: Use of the DSI/DA framework will change participants' knowledge about SCI and treatment options for people living with cervical SCI.
Decisional Conflict Questionnaire | At baseline and then immediately after reviewing the Decision Aid (estimated to be around 60-90 minutes later).
  An online questionnaire of 4 questions that are slightly modified, but based on the standardized, validated survey instrument called the SURE Test (of decisional conflict). This questionnaire will be administered as a "Pre-Test" before participants view the Decision Aid, and then later as a "Post-Test" after participants view the Decision Aid.
  Hypothesis: Participants will experience a change in decisional conflict when they think about improving arm and hand function in the setting of cervical spinal cord injury and consider the treatment options that they might prefer.

SECONDARY OUTCOMES:
Questionnaire to Assess the Acceptability of the Decision Aid | Immediately after reviewing the Decision Aid.
  An online questionnaire (14 questions) based on 3 standardized, validated survey instruments called the Acceptability Index, the System Usability Scale (SUS) and the Single Item Literacy Screener (SILS).They have been slightly modified for use in this population. This aggregated approach will provide information about the participant's experience with the Decision Aid and provide feedback on the overall helpfulness and suitability of the novel Decision Aid. The questionnaire will be administered as a "Post-Test" after participants view the Decision Aid.

CONTACTS AND LOCATIONS:
Overall Officials: Ida K Fox, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Nerve Transfers to Restore Upper Extremity Function in Cervical Spinal Cord Injury: Update and Preliminary Outcomes. Plast Reconstr Surg. 2015 Oct;136(4):780-792. doi: 10.1097/PRS.0000000000001641. PMID 26397252
- [Background] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Use of peripheral nerve transfers in tetraplegia: evaluation of feasibility and morbidity. Hand (N Y). 2015 Mar;10(1):60-7. doi: 10.1007/s11552-014-9677-z. PMID 25767422
- [Background] Curtin CM, Gater DR, Chung KC. Upper extremity reconstruction in the tetraplegic population, a national epidemiologic study. J Hand Surg Am. 2005 Jan;30(1):94-9. doi: 10.1016/j.jhsa.2004.10.007. PMID 15680562
- [Background] Bertelli JA, Ghizoni MF, Tacca CP. Transfer of the teres minor motor branch for triceps reinnervation in tetraplegia. J Neurosurg. 2011 May;114(5):1457-60. doi: 10.3171/2010.12.JNS101519. Epub 2011 Jan 21. PMID 21250798
- [Background] Bertelli JA, Ghizoni MF. Nerve transfers for elbow and finger extension reconstruction in midcervical spinal cord injuries. J Neurosurg. 2015 Jan;122(1):121-7. doi: 10.3171/2014.8.JNS14277. PMID 25343189
- [Background] Bertelli JA, Tacca CP, Ghizoni MF, Kechele PR, Santos MA. Transfer of supinator motor branches to the posterior interosseous nerve to reconstruct thumb and finger extension in tetraplegia: case report. J Hand Surg Am. 2010 Oct;35(10):1647-51. doi: 10.1016/j.jhsa.2010.07.012. PMID 20888500
- [Background] Friden J, Gohritz A. Brachialis-to-extensor carpi radialis longus selective nerve transfer to restore wrist extension in tetraplegia: case report. J Hand Surg Am. 2012 Aug;37(8):1606-8. doi: 10.1016/j.jhsa.2012.05.005. Epub 2012 Jun 30. PMID 22749482
- [Background] Curtin CM, Hayward RA, Kim HM, Gater DR, Chung KC. Physician perceptions of upper extremity reconstruction for the person with tetraplegia. J Hand Surg Am. 2005 Jan;30(1):87-93. doi: 10.1016/j.jhsa.2004.08.014. PMID 15680561
- [Background] Wagner JP, Curtin CM, Gater DR, Chung KC. Perceptions of people with tetraplegia regarding surgery to improve upper-extremity function. J Hand Surg Am. 2007 Apr;32(4):483-90. doi: 10.1016/j.jhsa.2007.01.015. PMID 17398358
- [Background] Fox PM, Suarez P, Hentz VR, Curtin CM. Access to surgical upper extremity care for people with tetraplegia: an international perspective. Spinal Cord. 2015 Apr;53(4):302-5. doi: 10.1038/sc.2015.3. Epub 2015 Feb 17. PMID 25687516
- [Background] Anderson KD, Friden J, Lieber RL. Acceptable benefits and risks associated with surgically improving arm function in individuals living with cervical spinal cord injury. Spinal Cord. 2009 Apr;47(4):334-8. doi: 10.1038/sc.2008.148. Epub 2008 Nov 25. PMID 19030014
- [Background] Cain SA, Gohritz A, Friden J, van Zyl N. Review of Upper Extremity Nerve Transfer in Cervical Spinal Cord Injury. J Brachial Plex Peripher Nerve Inj. 2015 Aug 6;10(1):e34-e42. doi: 10.1055/s-0035-1558427. eCollection 2015 Dec. PMID 27917237
- [Background] Joseph-Williams N, Newcombe R, Politi M, Durand MA, Sivell S, Stacey D, O'Connor A, Volk RJ, Edwards A, Bennett C, Pignone M, Thomson R, Elwyn G. Toward Minimum Standards for Certifying Patient Decision Aids: A Modified Delphi Consensus Process. Med Decis Making. 2014 Aug;34(6):699-710. doi: 10.1177/0272989X13501721. Epub 2013 Aug 20. PMID 23963501
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Mathers N, Ng CJ, Campbell MJ, Colwell B, Brown I, Bradley A. Clinical effectiveness of a patient decision aid to improve decision quality and glycaemic control in people with diabetes making treatment choices: a cluster randomised controlled trial (PANDAs) in general practice. BMJ Open. 2012 Nov 5;2(6):e001469. doi: 10.1136/bmjopen-2012-001469. Print 2012. PMID 23129571
- [Background] Barry MJ. Health decision aids to facilitate shared decision making in office practice. Ann Intern Med. 2002 Jan 15;136(2):127-35. doi: 10.7326/0003-4819-136-2-200201150-00010. PMID 11790064
- [Background] Volk RJ, Llewellyn-Thomas H, Stacey D, Elwyn G. Ten years of the International Patient Decision Aid Standards Collaboration: evolution of the core dimensions for assessing the quality of patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S1. doi: 10.1186/1472-6947-13-S2-S1. Epub 2013 Nov 29. PMID 24624947
- [Background] Coulter A, Stilwell D, Kryworuchko J, Mullen PD, Ng CJ, van der Weijden T. A systematic development process for patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S2. doi: 10.1186/1472-6947-13-S2-S2. Epub 2013 Nov 29. PMID 24625093
- [Background] Knops AM, Legemate DA, Goossens A, Bossuyt PM, Ubbink DT. Decision aids for patients facing a surgical treatment decision: a systematic review and meta-analysis. Ann Surg. 2013 May;257(5):860-6. doi: 10.1097/SLA.0b013e3182864fd6. PMID 23470574